CLINICAL TRIAL: NCT06023576
Title: Intensive Blood Pressure Control During Cardiotoxic Breast Cancer Treatment (PROTECT), A Randomized Controlled Trial
Brief Title: A Study of Blood Pressure Control During Cancer Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-159
Record Dates: First submitted 2023-08-18; First posted 2023-09-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Cardiotoxicity
Keywords: Blood pressure; 23-159
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Blood Pressure Determination; Echocardiography; Environmental Biomarkers

STUDY DESIGN:
Intervention Model Description: This open-label, two-arm RCT will compare the effects of intensive versus standard SBP control in patients with BC and HTN receiving anthracycline-based treatment (with or without HER2-targeted therapy).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard-of-care antihypertensive medications (Experimental): SBP control will consist of treatment with antihypertensive medications titrated every 4 weeks for the first 3 months, and then every 3 months in months 4-12. SBP control will be achieved by titration of antihypertensive medications based upon a standardized algorithm and will be implemented during a 12-month study period. At the time of randomization, no antihypertensive treatments may be initiated or modified if SBP is ≥160 mm Hg. The clinical context may be considered at each visit to inform decision-making regarding treatment initiation or modification, at the discretion of the treating provider.
  Interventions: Other: antihypertensive medications; Diagnostic Test: Blood pressure measurement; Diagnostic Test: Echocardiogram; Other: Symptom-limited cardiopulmonary exercise test; Other: Quality of Life Measures; Diagnostic Test: Biomarkers
- higher dose antihypertensive medications (Experimental): Patients randomized to intensive SBP control will be treated to achieve an SBP goal <120 mm Hg, and patients randomized to standard SBP control will be treated to achieve an SBP goal <140 mm Hg. Antihypertensive medications will be titrated on the basis of seated blood pressure measurements obtained after a 5-min rest period. All participants will be provided with dietary (e.g., 1500mg/d sodium restriction) and lifestyle recommendations as background therapy for optimizing HTN control.The clinical context may be considered at each visit to inform decision-making regarding treatment initiation or modification, at the discretion of the treating provider.
  Interventions: Other: antihypertensive medications; Diagnostic Test: Blood pressure measurement; Diagnostic Test: Echocardiogram; Other: Symptom-limited cardiopulmonary exercise test; Other: Quality of Life Measures; Diagnostic Test: Biomarkers

INTERVENTIONS:
Other: antihypertensive medications — One or more of the following medications may be used in both randomization groups to achieve SBP goals:
  * Angiotensin converting enzyme inhibitors (ACEI)
  * Angiotensin receptor blockers (ARBs)
  * Beta-blockers (BB)
  * Thiazide-type diuretics
  * Calcium channel blockers
  * Aldosterone antagonists
  * Alpha1-receptor blockers.
  * Direct vasodilators
  * Loop diuretics
Diagnostic Test: Blood pressure measurement — Home BP Monitoring (HBPM)-Throughout the study period, patients will perform HBPM at baseline, month 6, and month 12 (end of treatment). At each of these timepoints, HBPM will be performed for 7 days with 2 morning and 2 evening readings for each day (measured 1-min part).
Diagnostic Test: Echocardiogram — At baseline, month 6, and month 12
Other: Symptom-limited cardiopulmonary exercise test — Consecutive patients in each treatment group who meet the eligibility criteria for exercise testing will be offered to participate in CPET at the time of consent. Patients who agree will undergo CPET (baseline, 6 months, and 12 months) until the target accrual of 33 patients per group is met.
Other: Quality of Life Measures — FACT-B, Fatigue Symptom Inventory (FSI), Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale, Godin Leisure Time Exercise Questionnaire (GLTEQ),PROMIS Medication Adherence Scale. Given baseline, 3 months and 12 months.
Diagnostic Test: Biomarkers — Research blood samples will be collected at baseline, 3 months, and 6 months

SUMMARY:
The purpose of this study to find out whether an intensive approach to treating high blood pressure during breast cancer treatment is safe and more effective than standard blood pressure treatment at lowering blood pressure levels and the risk of cardiotoxicity in patients with cancer. Other studies have shown lowering blood pressure improves the health of patients. However, these studies have not included people with cancer.

The PROTECT trial is testing a treatment strategy regarding intensive versus standard SBP goals, and is not testing specific medications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Female assigned at birth
* Biopsy proven breast cancer (stage I-IV)
* Treatment with therapy anthracycline-based chemo (with or without HER2-targeted therapy), with >/= 2 cycles of anthracycline chemotherapy planned.
* SBP ≥130 mm Hg
* Willing and able to comply with the requirements of the protocol.
* Participant must have and be willing to use their bluetooth enabled wifi or cellular mobile device
* (For participants in the CPET cohort): Able to complete an acceptable baseline CPET, in the absence of high-risk ECG findings or other inappropriate response to exercise as determined by the PI, as defined by any of the following criteria:

  * Achieving a plateau oxygen consumption, concurrent with an increase in power output;
  * A respiratory exchange ratio ≥ 1.10;
  * Attainment of maximal predicted heart rate, as defined by a peak heart rate within 10bpm of the age predicted maximal heart rate (220 - Age[years]);
  * Volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale.

Exclusion Criteria:

* eGFR < 30 ml/min/1.73m2 (based upon Cockcroft-Gault, etc.)
* Individuals with arm circumference too large to allow accurate BP measurement with available BP devices
* Inability to accurately measure blood pressure in at least one arm (e.g., bilateral upper extremity lymphedema)
* Cardiac comorbidity, including any of the following:

  * Acute coronary syndrome within 3 months prior to randomization.
  * Symptomatic heart failure (NYHA class III/IV) within past 6 months
  * History of stroke
  * Cardiac transplantation
* Other medical disorder or condition that in the opinion of the investigator would impair the subject's ability to participate or adhere to study interventions
* (For participants in the CPET cohort): Subjects must not have any of the following absolute contraindications to cardiopulmonary exercise testing:

  * Acute myocardial infarction (within 30 days of any planned study procedures),
  * Unstable angina
  * Uncontrolled arrhythmias causing symptoms or hemodynamic compromise,
  * Symptomatic severe aortic stenosis
  * Recurrent syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Acute pulmonary embolus or pulmonary infarction (within 3 months of any planned study procedures)
  * Thrombosis of lower extremities (within 3 months of any planned study procedures)
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Pulmonary edema
  * Room air desaturation at rest ≤85%
  * Respiratory failure
  * Acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis)
  * Mental impairment leading to inability to cooperate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female assigned at birth
Enrollment: 130 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
mean change in systolic blood pressure (SBP) from baseline to 12 months | 12 months
  based upon in-office measurement

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm